CLINICAL TRIAL: NCT04680195
Title: Prospective, Open Clinical Trial of Thalidomide in the Treatment of Chronic Radiation Proctitis With Intractable Bleeding
Brief Title: Thalidomide in the Treatment of Chronic Radiation Proctitis With Intractable Bleeding
Acronym: Thal-CRP
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Sixth Affiliated Hospital, Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HOPE2020-Thal-CRP
Record Dates: First submitted 2020-12-02; First posted 2020-12-22 (Actual); Last update posted 2020-12-22 (Actual); Status verified 2020-12

CONDITIONS: Chronic Radiation Proctitis
Keywords: Thalidomide; Bleeding; Chronic radiation proctitis
MeSH Terms: conditions — Hemorrhage | interventions — Thalidomide

STUDY DESIGN:
Intervention Model Description: Thalidomide Group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Thalidomide treatment Group (Experimental): Induction period:
  Thalidomide tablets: 50-100 mg/d, qn, po.
  Maintenance period:
  Thalidomide tablets: 50-75 mg/d qn, po.
  Interventions: Drug: Thalidomide

INTERVENTIONS:
Drug: Thalidomide — The patients were treated with thalidomide tanken orally every night for 4 months, and the treatment period was divided into induction period and maintenance period, as follows:
  Induction period:
  The oral dose of thalidomide started at 50 mg, and increased to 100 mg after one week if tolerable, and maintain 100 mg for three weeks. The medication time was 1 month.
  Maintenance period: The oral dose of thalidomide was 50-75mg/d. The medication time was 3 months.

SUMMARY:
Chronic radiation proctitis (CRP) is the main secondary toxic injury after pelvic radiotherapy. Hematochezia is the most common symptom for more than 80% of CRP patients.

Non-surgical treatment is the first choice to the treatment of CRP to avoid the occurrence of serious complications. Conventional oral medication for the treatment of bleeding CRP is very few and has little effect. At present, no oral medication has been found to significantly alleviate and control refractory bleeding of CRP. Therefore, it is an urgent problem to screen out a drug that is more effective, safe and highly compliant for the treatment of hemorrhagic CRP.

Thalidomide has anti-inflammatory, immune regulation, anti-angiogenesis and other effects. For the patients of CRP with intractable bleeding, a prospective, open clinical trial will be carried out to observe the safety and effectiveness of thalidomide in treating hemorrhagic CRP.

DETAILED DESCRIPTION:
Radiotherapy is an essential therapeutic tool for pelvic malignancies such as uterine cervix, uterine corpus, prostate, testicular, urinary bladder and rectal cancers. According to reports, the estimated number of new cases of malignant pelvic tumors in China in 2015 alone exceeded 500,000. Chronic radiation proctitis (CRP) is an unavoidable and commonly observed side effect, occurs 3 months later and in 5-20% of patients after pelvic malignancy radiation. Hematochezia is the most common symptom for more than 80% of CRP patients, which is a persistent, irreversible and progressive symptom, and will probably give rise to anemia. In clinic, the treatment for intractable bleeding of CRP is very difficult.

Non-surgical treatment is the first choice to the treatment of CRP to avoid the occurrence of serious complications. Conventional oral medication for the treatment of bleeding CRP is very few and has little effect. At present, no oral medication has been found to significantly alleviate and control refractory bleeding of CRP. Therefore, it is an urgent problem to screen out a drug that is more effective, safe and highly compliant for the treatment of hemorrhagic CRP.

Thalidomide has anti-inflammatory, immune regulation, anti-angiogenesis and other effects. A large number of studies have shown that thalidomide can be used to treat Crohn's disease, ulcerative colitis, radiation cystitis, etc., and it can treat moderate to severe of IBD patients can inhibit inflammatory response, improve clinical symptoms, promote intestinal mucosal repair. Further, recent studies have proved that thalidomide can be used to treat intestinal bleeding due to vascular dysplasia. And a case report from Gut described that refractory bleeding of CRP of a 78-year-old woman were significantly alleviated after taking thalidomide.

Therefore, for the patients of CRP with intractable bleeding, a prospective, open clinical trial planed to carry out to observe the safety and effectiveness of thalidomide in treating hemorrhagic CRP.

ELIGIBILITY:
Inclusion criteria

1. Patients aged 18-75 years;
2. Patients with ECOG physical condition score of 0-2;
3. Patients with previous pathological diagnosis of pelvic tumors (Gynecology, prostate, urinary system);
4. Patients with a history of pelvic radiotherapy, at least 6 months from the end of the last radiotherapy;
5. Patients with no primary tumor recurrence or metastasis;
6. Patients with refractory hemorrhagic CRP who have failed to conventional treatment (SOMA score for hematochezia≥2, hemoglobin level ≤90g/L, or a history of blood transfusion due to CRP)
7. Subjects and their family members can understand the research plan, and are willing to participate, and sign an informed consent form.

Exclusion Criteria:

1. Patients with active bleeding requiring emergency treatment;
2. Patients with severe complications of CRP, such as Rectal ulcer (VRS>Grade 3) or fistula, perforation, stenosis, necrosis, perianal intractable pain and so on
3. Patients with a history of rectal resection;
4. Other bleeding diseases, such as grade III or IV hemorrhoids, coagulation dysfunction, etc.;
5. Patients with other diseases requiring long-term use of anticoagulant drugs;
6. Combined intestinal obstruction, requiring surgery;
7. The absolute value of neutrophils of patients is lower than 750/mm3;
8. Patients who are allergic to thalidomide;
9. Pregnant or lactating women;
10. Patients with severe mental illness;
11. Patients who cannot take medication or follow up as planned;
12. During the trial and within 3 months after the trial, the subjects and their partners are not willing to contraception;
13. Participants in other clinical investigators 3 months before the trial

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2020-12-14 (Estimated); Primary Completion 2022-07-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
Remission rate of rectal bleeding one month after thalidomide treatment | the first month after thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.

SECONDARY OUTCOMES:
Remission rate of rectal bleeding one month during thalidomide treatment | the first month during thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Remission rate of rectal bleeding two months during thalidomide treatment | the second month during thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Remission rate of rectal bleeding three months during thalidomide treatment | the third month during thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Remission rate of rectal bleeding four months during thalidomide treatment | the fourth month during thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Remission rate of rectal bleeding three months after thalidomide treatment | the third month after thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Remission rate of rectal bleeding six months after thalidomide treatment | the sixth month after thalidomide treatment
  Remission of rectal bleeding was defined as the score of Subjective Objective Management Analysis system (SOMA) for retcal bleeding at least 1 grade lower and the hemoglobin level at least 10g/L higher than that before treatment. The SOMA score for hematochezia was ranged from 1 to 4, with the higher the score, the more serious.
Endoscopic score one month during thalidomide treatment | the first month during thalidomide treatment
  Endoscopic score was performed using Vienna rectoscopy Score (VRS). VRS was ranged 1 to 5. A higher score indicated a more severe lesion.
Endoscopic score four months during thalidomide treatment | the fourth month during thalidomide treatment
  Endoscopic score was performed using Vienna rectoscopy Score (VRS). VRS was ranged 1 to 5. A higher score indicated a more severe lesion.
Endoscopic score one month after thalidomide treatment | the first month after thalidomide treatment
  Endoscopic score was performed using Vienna rectoscopy Score (VRS). VRS was ranged 1 to 5. A higher score indicated a more severe lesion.
Endoscopic score three months after thalidomide treatment | the third month after thalidomide treatment
  Endoscopic score was performed using Vienna rectoscopy Score (VRS). VRS was ranged 1 to 5. A higher score indicated a more severe lesion.
Endoscopic score six months after thalidomide treatment | the sixth month after thalidomide treatment
  Endoscopic score was performed using Vienna rectoscopy Score (VRS). VRS was ranged 1 to 5. A higher score indicated a more severe lesion.
Quality of life of the patient one month during thalidomide treatment | the first month during thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 is a 30-item questionnaire composed of multi-item scales and single items that reflect the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient two months during thalidomide treatment | the second month during thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient three months during thalidomide treatment | the third month during thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient four months during thalidomide treatment | the fourth month during thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient one month after thalidomide treatment | the first month after thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient three months after thalidomide treatment | the third month after thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Quality of life of the patient six months after thalidomide treatment | the sixth month after thalidomide treatment
  Quality of life of the patient was evaluated by the European Organisation for the Research and Treatment of Cancer Quality of Life Questionnaire Core 30 (EORTC QLQ-C30). The EORTC QLQ-C30 was a 30-item questionnaire composed of multi-item scales and single items that reflecting the multidimensionality of the quality-of-life. It incorporated five functioning subscales (physical, role, cognitive, emotional, and social), nine symptom subscales (pain, fatigue, nausea and vomiting, appetite loss, constipation, diarrhea, dyspnea, insomnia, financial difficulties), and one global quality of life subscale, and the scores were ranged 0 to 100. Higher scores for functional subscales and global quality of life subscale indicated the better functional status and quality of life. But the higher scores for symptom subscales indicated the poorer quality of life.
Incidence of adverse events four months during thalidomide treatment | the fourth month during thalidomide treatment
  Including adverse reactions of thalidomide and other adverse events
Incidence of adverse events six months after thalidomide treatment | the sixth month after thalidomide treatment
  Including adverse reactions of thalidomide and other adverse events

REFERENCES:
- [Background] Yuan ZX, Ma TH, Zhong QH, Wang HM, Yu XH, Qin QY, Chu LL, Wang L, Wang JP. Novel and Effective Almagate Enema for Hemorrhagic Chronic Radiation Proctitis and Risk Factors for Fistula Development. Asian Pac J Cancer Prev. 2016;17(2):631-8. doi: 10.7314/apjcp.2016.17.2.631. PMID 26925655
- [Background] Andreyev HJ. Argon plasma coagulation in chronic radiation proctitis: Postgate et al. Endoscopy. 2007 Aug;39(8):751-2; author reply 752. doi: 10.1055/s-2007-966772. No abstract available. PMID 17661253
- [Result] Craanen ME, van Triest B, Verheijen RH, Mulder CJ. Thalidomide in refractory haemorrhagic radiation induced proctitis. Gut. 2006 Sep;55(9):1371-2. doi: 10.1136/gut.2006.099416. No abstract available. PMID 16905712
- [Result] Zhou S, Wang F, Hsieh TC, Wu JM, Wu E. Thalidomide-a notorious sedative to a wonder anticancer drug. Curr Med Chem. 2013;20(33):4102-8. doi: 10.2174/09298673113209990198. PMID 23931282
- [Result] Yuan ZX, Ma TH, Wang HM, Zhong QH, Yu XH, Qin QY, Wang JP, Wang L. Colostomy is a simple and effective procedure for severe chronic radiation proctitis. World J Gastroenterol. 2016 Jun 28;22(24):5598-608. doi: 10.3748/wjg.v22.i24.5598. PMID 27350738
- [Result] Kim KT, Chae HS, Kim JS, Kim HK, Cho YS, Choi W, Choi KY, Rho SY, Kang SJ. Thalidomide effect in endothelial cell of acute radiation proctitis. World J Gastroenterol. 2008 Aug 14;14(30):4779-83. doi: 10.3748/wjg.14.4779. PMID 18720539
- [Result] Bauditz J, Wedel S, Lochs H. Thalidomide reduces tumour necrosis factor alpha and interleukin 12 production in patients with chronic active Crohn's disease. Gut. 2002 Feb;50(2):196-200. doi: 10.1136/gut.50.2.196. PMID 11788559
- [Result] Alberto SF, Felix J, de Deus J. Thalidomide for the treatment of severe intestinal bleeding. Endoscopy. 2008 Sep;40(9):788; author reply 789. doi: 10.1055/s-2008-1077513. Epub 2008 Sep 4. No abstract available. PMID 18773348
- [Result] Bauditz J, Schachschal G, Wedel S, Lochs H. Thalidomide for treatment of severe intestinal bleeding. Gut. 2004 Apr;53(4):609-12. doi: 10.1136/gut.2003.029710. PMID 15016759
- [Result] McCrone LF, Neary PM, Larkin J, McCormick P, Mehigan B. The surgical management of radiation proctopathy. Int J Colorectal Dis. 2017 Aug;32(8):1099-1108. doi: 10.1007/s00384-017-2803-y. Epub 2017 Apr 20. PMID 28429071
- [Result] Ma TH, Yuan ZX, Zhong QH, Wang HM, Qin QY, Chen XX, Wang JP, Wang L. Formalin irrigation for hemorrhagic chronic radiation proctitis. World J Gastroenterol. 2015 Mar 28;21(12):3593-8. doi: 10.3748/wjg.v21.i12.3593. PMID 25834325